CLINICAL TRIAL: NCT04965610
Title: Preoxygenation With High Flow Nasal Cannula Prolongs Normoxia Time During Induction of Anaesthesia of Bariatric Patients and is Superior to Conventional Preoxygenation With Face Mask.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Staedtisches Klinikum Karlsruhe (Other)
Responsible Party: Principal Investigator, Joachim Jugl, Assistenzarzt Anästhesie, Staedtisches Klinikum Karlsruhe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 070720211
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Compare Preoxygenation Methods in Bariatric Patients

STUDY DESIGN:
Intervention Model Description: Two groups of patients. One receiving preoxygenation via High Flow Nasal Cannula and one group receiving preoxygenation via face mask
Masking Description: Patients will be divided into two groups by lot.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoxygenation via THRIVE/High Flow Nasal Cannula (Experimental): Patients receive preoxygenation for induction of general anaesthesia via High Flow Nasal Cannula for the duration of 5 minutes. After that the induction agents will be given. Now arterial blood gases will be drawn every 2 minutes and the SpO2 will be measured until the 6th apnoeic ABG or if the SpO2 decreases to 92%. After that normal intubation follows.
  Interventions: Other: Preoxygenation with High Flow Nasal Cannula
- Preoxygenation via face mask (PROX) (Active Comparator): Patients receive preoxygenation for induction of general anaesthesia via tight fitting face mask for the duration of 5 minutes. After that the induction agents will be given. Now arterial blood gases will be drawn every 2 minutes and the SpO2 will be measured until the 6th apnoeic ABG or if the SpO2 decreases to 92%. After that normal intubation follows.
  Interventions: Other: Preoxygenation via face mask

INTERVENTIONS:
Other: Preoxygenation with High Flow Nasal Cannula — Preoxygenation for 5 minutes via High Flow Nasal Cannula. After induction of anaesthesia apnoeic oxygenation with HFNC
  Arms: Preoxygenation via THRIVE/High Flow Nasal Cannula
Other: Preoxygenation via face mask — Preoxygenation for 5 minutes via face mask. After induction of anaesthesia apnoeic oxygenation with tight fitting face mask
  Arms: Preoxygenation via face mask (PROX)

SUMMARY:
To compare preoxygenation for induction of general anaesthesia with High Flow Nasal Cannula vs preoxygenation with face mask in patients undergoing bariatric surgery. The hypothesis is that preoxygenation with High Flow Nasal Cannula prolongs normoxia time during induction of anaeshesia and is superior to conventional preoxygenation with face mask. Primary endpoint will be the time during which spO2 > 92 %. Secondary endpoint will be paCO2.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* elective bariatric surgery
* written consent

Exclusion Criteria:

* preexisting lung diseases, congenital heart diseases
* known difficult airway
* SpO2 < 92% under ambient air conditions
* known diaphragmal hernia
* clinically relevant reflux

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Normoxia time SpO2 > 92% | 10 Minutes after induction
  Time in which the SpO2 remains > 92% while patient is apnoeic

SECONDARY OUTCOMES:
paCO2 | 10 Minutes after induction
  Increase in arterial CO2 during Apnoea

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Jugl, Principal Investigator — Senior Resident Anaesthesia; Franz Kehl, Prof., Study Director — Head of Department of Anaesthesia and Intensive Care

IPD SHARING:
Plan to Share IPD: Undecided